CLINICAL TRIAL: NCT05414136
Title: A Single-arm, Open, Dose-increasing Phase I Clinical Study Evaluating the Safety, Tolerability, and Pharmacokinetics of BAT1006 in Patients with Her2-positive Advanced Solid Tumors
Brief Title: Evaluating the Safety, Tolerability, and Pharmacokinetics of BAT1006
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-1006-001-CR
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- A1/3mg/kg (Experimental): Dose: 3mg/kg
  Interventions: Drug: BAT1006
- A2/6mg/kg (Experimental): Dose: 6mg/kg
  Interventions: Drug: BAT1006
- A3/10mg/kg (Experimental): Dose: 10mg/kg
  Interventions: Drug: BAT1006
- A4/15mg/kg (Experimental): Dose: 15mg/kg
  Interventions: Drug: BAT1006
- A5/20mg/kg (Experimental): Dose: 20mg/kg
  Interventions: Drug: BAT1006

INTERVENTIONS:
Drug: BAT1006 — Intravenous fluids
  Other Names: Recombinant humanized anti-HER2 monoclonal antibody for injection

SUMMARY:
Primary objectives: To evaluate the safety and tolerability of BAT1006 in patients with advanced her2-positive solid tumors. To determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT).

Secondary objectives: 1) To evaluate the pharmacokinetic characteristics of BAT1006 after single and multiple dosing; 2) To study the immunogenicity of BAT1006; 3) Preliminary evaluation of anti-tumor efficacy of BAT1006.

DETAILED DESCRIPTION:
This trial is an open phase I, dose-escalation clinical study. The first administration period was the 21st day, namely the DLT observation period. DLT observation was conducted to explore the safety, tolerability, pharmacokinetics and immunogenicity of MTD, single administration. After the observation period of DLT, the drug was administered once every 3 weeks, and the tolerance, pharmacokinetics, immunogenicity and preliminary effectiveness of multiple administration were evaluated. If some dose groups show better efficacy, the investigator and the sponsor may select 1-2 dose groups that have been found to have efficacy after negotiation and discussion for extended study to further explore the safety and efficacy of the drug.

ELIGIBILITY:
inclusion criteria：

1. The patient or his legal representative signs the informed consent, fully understands the content, process and possible adverse reactions of the trial, and is willing to conduct follow-up and imaging evaluation in accordance with the time specified in the trial;
2. Age 18-80 years old (including boundary value), gender is not limited;
3. Patients with locally advanced or metastatic solid tumors confirmed by histopathology and/or cytology as HER2-positive. The extended study was limited to patients with HER2-positive locally advanced or metastatic breast and stomach cancer. Her2-positive (HER2-positive defined as IHC3+ or FISH+);
4. Patients with no effective treatment or failure of standard treatment;
5. Tumor with at least one measurable lesion according to Recist version 1.1 criteria;
6. United States Eastern Oncology Collaboration (ECOG) physical status score 0-1;
7. Expected survival ≥3 months;
8. Have sufficient bone marrow, liver, kidney and blood clotting function,
9. Left ventricular ejection fraction (LVEF) ≥55% by echocardiography;
10. Fertile female patients must have a negative serological pregnancy test prior to first dosing and be willing to use an effective birth control/contraceptive method to prevent pregnancy during the study period up to 6 months after the last dosing of the study. Male patients must consent to an effective contraceptive method for the duration of the study up to 6 months after the last dosing in the study.

exclusion criteria:

1. Previous doxorubicin cumulative dose > Subjects with 360 mg/m2 or equivalent anthracyclines;
2. Previous treatment with trastuzumab, pertuzumab, or other HER2-targeted drugs (including but not limited to grade 3 or higher infusion reactions or allergic reactions, LVEF < 50% after treatment, or grade 3 or higher diarrhea);
3. The toxic effects of previous antitumor therapy have not returned to grade 0 to 1 as defined in CTCAE version 5.0, except for alopecia, pigmentation and anemia;
4. Patients who have received other anti-tumor therapy, such as chemotherapy, radiotherapy (but for palliative radiotherapy within 2 weeks before the first dose), biological products, etc., within 4 weeks of the first dose (targeted therapy/immunotherapy with a minimum interval of 4 weeks or at least 5 half-lives, whichever is shorter; Within 6 weeks before administration of nitrosourea and mitomycin C, within 2 weeks before administration of oral fluorouracil, within 1 week before administration of NMPA-approved Chinese patent medicine or treatment clearly with anti-tumor related functions, or Chinese herbal therapy clearly recorded in the medical records for anti-tumor purposes);
5. The presence of ≥2 grade peripheral neuropathy (CTCAE5.0 grade);
6. Pregnant or nursing women;
7. Patients with CNS metastases that are symptomatic or require ongoing treatment, but asymptomatic and radiologically stable for more than 4 weeks without the need for corticosteroid treatment could be enrolled;
8. Patients with active infection prior to initial administration and currently in need of intravenous anti-infective therapy;
9. Patients infected with any of the following viruses: active hepatitis B (HBsAg (+), with HBV DNA > 500IU/ml or the maximum hospital limit); Active hepatitis C (HCV antibody positive and HCV-RNA levels above the lower limit of detection); HIV infection; Active syphilis infection (RPR positive);
10. Have active pneumonia/interstitial lung disease (ILD), a history of pneumonia/interstitial lung disease requiring systemic steroid treatment, have received lung radiation within 12 months prior to the first administration of the study drug, or currently have clinically relevant lung disease (such as chronic obstructive pulmonary disease);
11. Active autoimmune diseases requiring systemic treatment (such as the use of disease-regulating drugs, corticosteroids, or immunosuppressive drugs), allowing for relevant replacement therapy (such as thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency);
12. Serious signs and symptoms accompanied by other concurrent, severe, or uncontrollable systemic diseases, including but not limited to: active gastric ulcers, uncontrolled epilepsy, cerebrovascular accidents, gastrointestinal bleeding, blood clotting and coagulation disorders;
13. Cardiovascular abnormalities within the first 6 months of enrollment according to any of the following definitions: Based on the CTCAE5.0 standard grade ≥3 symptomatic congestive heart failure (CHF), or the New York Heart Society (NYHA) standard grade ≥2 symptomatic congestive heart failure, transmastic myocardial infarction, and unstable angina pectoris, Or severe arrhythmia, severe conduction block, poorly controlled hypertension (blood pressure after medication > 150/100 MMHG), or other clinically significant cardiovascular disease;
14. Have participated in and received other clinical trials within 4 weeks before the first dose;
15. Received any live virus vaccine within 4 weeks prior to the first dose;
16. Have received major surgical treatment within 4 weeks prior to the first dose and have not fully recovered;
17. Known or suspected allergy to test drug components;
18. Researchers believe that participants are not suitable for this experiment for other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 21 days
  Dose-limiting toxicity (DLT) is defined as any of the following adverse events (CTCAE Version 5.0 classification for the evaluation of adverse effects) that occur during the first treatment cycle that are definitely or possibly related to the investigatory drug:
  1. Grade ≥3 non-hematological toxicity (nausea, vomiting and diarrhea can be relieved within 3 days after supportive treatment, except for infusion reactions that can be recovered within 2 hours after symptomatic treatment);
  2. Hematological toxicity 2.1 Grade ≥3 neutropenia with fever, or grade 3 thrombocytopenia with significant bleeding; 2.2 Grade ≥4 hematologic toxicity: thrombocytopenia for more than 5 days, or grade 4 neutropenia for more than 7 days;
  3. LVEF decreased by > 15% or LVEF value decreased by < 50% from baseline;
  4. In the case of other SAE or AE that the researcher considers unacceptable, the researcher will communicate with the sponsor to decide whether to judge it as DLT.
Maximum tolerance dose（MTD） | 21 days
  MTD is defined as the highest dose level of DLT observed in ≤1/6 subjects in a dose group during the DLT evaluation period

CONTACTS AND LOCATIONS:
Overall Officials: Shusen Wang, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No